CLINICAL TRIAL: NCT05216913
Title: Optimising Cardiovascular Health in Endometrial Cancer Survivors
Acronym: OPTIMUS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Emma Crosbie, Professor, University of Manchester
Other Study IDs: IRAS 298610
Record Dates: First submitted 2022-01-04; First posted 2022-02-01 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Endometrial Cancer; Cardiovascular Diseases
MeSH Terms: conditions — Endometrial Neoplasms; Cardiovascular Diseases | interventions — Cardiovascular Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endometrial cancer survivors
  Interventions: Behavioral: Lifestyle modification; Drug: Cardiovascular Agents, Other; Other: QRISK 3 Score

INTERVENTIONS:
Behavioral: Lifestyle modification — Could include all/some of the following: weight loss, increased physical activity, smoking cessation and reduction in alcohol intake
Drug: Cardiovascular Agents, Other — Could include all/some of the following: statins, antihypertensives, diabetic medication, levothyroxine
Other: QRISK 3 Score — Could include a combination of lifestyle measures and/or cardiovascular agents as described above

SUMMARY:
Women successfully treated for endometrial cancer remain at higher risk of dying than women without a history of the disease, predominately due to an excess risk of cardiovascular disease. Our previous work has shown that endometrial cancer survivors are more likely to have undiagnosed and undertreated cardiovascular risk factors than the general population, despite being seen regularly by medical professionals. This study aims to determine the impact of optimising modifiable cardiovascular risk factors in endometrial cancer survivors on their quality of life and to identify barriers to lifestyle modifications.

DETAILED DESCRIPTION:
A comprehensive cardiovascular risk assessment will be performed as part of clinical care on women previously treated for endometrial cancer at the study site. This will include a focused interview, examination to determine body mass index (BMI) and waist circumference, blood pressure, blood tests and a urine sample.

The blood tests will screen for diabetes and non-diabetic hyperglycaemia (HbA1c), renal impairment (full blood count- FBC, urea and electrolytes- U&E), non-alcoholic fatty liver disease and contraindication to statin therapy (liver function tests- LFT), hypercholesterolaemia (total, HDL and LDL cholesterol) and hypothyroidism (thyroid function tests- TFT). Urine samples will be used to screen for renal impairment using dipstick testing for microscopic haematuria and determination of albumin: creatinine ratio (ACR).

An individualised cardiovascular risk assessment will be undertaken using the QRISK3 score, which is assessed by virtue of the presence or absence of individual cardiovascular risk factors.

Based on these findings, an individualised management plan will be generated and appropriate treatment for any modifiable risk factors commenced in accordance with NICE (National Institute for Health and Care Excellence) and local guidelines. This will include advice and support with lifestyle modification, commencing medication if needed and referral to community or specialist clinics. This will be carried with close communication and in conjunction with the patient's general practitioner (GP).

Women will be followed up over a one year period to monitor their response and compliance to treatment and the impact this has on their quality of life.

The quality of life assessments will be undertaken by a member of the research team using the generic 36-Item Short Form Survey [SF-36] and cancer-specific Quality of Life in Adult Cancer Survivors [QLACS] questionnaires. A subset of approximately twenty women, purposively sampled to include maximal variation in age, body mass index and time from diagnosis, will be selected to participate in a qualitative study of the barriers to the implementation and adherence of lifestyle interventions.

Study visits will be timed to coincide with routine follow-up appointments or be carried out remotely by telephone or Zoom to minimise the risk of COVID-19 exposure. Follow-up visits will consist of a focused interview and quality of life questionnaires, with a repeat of the comprehensive cardiovascular risk assessment at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Previous treatment for endometrial cancer within the last four years
* Able to consent to participation in the study

Exclusion Criteria:

* Currently undergoing treatment for endometrial cancer recurrence
* Anticipated life expectancy <12 months
* To cease routine surveillance in next 12 months
* Not registered with a General Practitioner (GP)

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who have had endometrial cancer treated within the last 4 years.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
To assess the change in quality of life in endometrial cancer survivors by treating modifiable cardiovascular risk factors over a period of 12 months. | Baseline, 3 months, 6 months and 12 months.
  The generic 36-Item Short Form Survey (SF-36) questionnaire focused on general wellbeing and quality of life.
  A variety of responses are used in this questionnaire. Some use numeric indicators, with a lower overall score meaning a worse outcome and a higher score meaning a better outcome.
To assess the change in quality of life in endometrial cancer survivors by treating modifiable cardiovascular risk factors over a period of 12 months. | Baseline, 3 months, 6 months and 12 months.
  The cancer-specific Quality of Life in Adult Cancer Survivors (QLACS) questionnaire focused on general well-being and quality of life.
  This questionnaire uses numeric indicators from 1 to 7, with a lower overall score meaning a worse outcome and a higher score meaning a better outcome.

SECONDARY OUTCOMES:
To identify barriers to the implementation of lifestyle changes in endometrial cancer survivors. | Between 3 and 9 months.
  A subset of approximately twenty women, will take part in semi-structured interviews to discuss barriers to implementation and adherence to lifestyle interventions. Questioning will focus on the motivations, opportunities and capability of individuals to change their behaviour and will be thematically analysed, with particular attention paid to features of the Behavioural Change Wheel.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Crosbie, Principal Investigator — University of Manchester
Locations (1):
- St Mary's Hospital, Manchester, United Kingdom